CLINICAL TRIAL: NCT03808181
Title: An Open, Single-arm, Multi Centre Pilot Investigation to Evaluate the Debriding Effect of ChloraSolv® on Chronic Wounds, Covered With Devitalised Tissue, During Six Weeks Treatment
Brief Title: An Open, Single-arm, Multi Centre Pilot Investigation to Evaluate the Debriding Effect of ChloraSolv® on Chronic Wounds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RLS Global (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ChloraSolv 01
Record Dates: First submitted 2019-01-14; First posted 2019-01-17 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Chronic Ulcer at Lower Leg

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Active treatment with ChloraSolv (Other): Single arm
  Interventions: Device: ChloraSolv

INTERVENTIONS:
Device: ChloraSolv — Weekly application of ChloraSolv for 6 weeks

SUMMARY:
The primary objective of this clinical investigation is to evaluate the debriding effect of ChloraSolv® on chronic (more than 1 moth) lower leg ulcer.

DETAILED DESCRIPTION:
Approximately 58 subjects from at least two sites in Sweden will be included. Subjects presented with lower leg ulcer, covered with devitalised tissue for 50% or more and being candidate for cleansing, debridement/desloughing will be enrolled. Weekly application of Investigational Product for 6 weeks. Follow-up for wound status evaluation after 12 weeks from baseline. Total time in investigation is 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Full skin ulcer at lower leg covered with devitalised tissue ≥50%
2. Candidate for cleansing, debridement/desloughing
3. Wound area ≥2 cm²
4. Male or female, 18 years of age and above
5. Able to read and understand the Patient Informed Consent and to provide meaningful written informed consent
6. Able and willing to follow the Protocol requirements

Exclusion Criteria:

1. Clinical signs of system progression infection with or without ostemyelitis
2. Wound located where treatment is not possible
3. Subjects not suitable for the investigation according to the investigator's judgment
4. Subjects included in other ongoing clinical investigation which could interfere with this investigation, as judged by the investigator
5. Known allergy/hypersensitivity to any of the components of the investigational device
6. Pregnant or breast feeding women
7. Other significant medical condition that the investigator determines could interfere with compliance or study assessments
8. Subjects with wounds of duration less than one month
9. Wound area greater than approximately 60 cm²

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2019-01-31 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
The primary objective of this clinical investigation is to evaluate the debriding effect of ChloraSolv® on chronic (more than 1 month) lower leg ulcer. | 6 weeks
  The debriding effect of ChloraSolv® will be assessed by planimetry (photography) prior to and after each debridement. The photos will be sent for evaluation by an independent assessor.

SECONDARY OUTCOMES:
The secondary objectives are to evaluate change of devitalised tissue, change in wound area, pain during treatment, condition of the wound, need for sharp debridement and overall evaluation of the product and safety parameters. | 12 weeks
  The objectives to evaluate change of devitalised tissue and change in wound area will be assessed by planimetry (photography) prior to and after each debridement. The photos will be sent for evaluation by an independent assessor. Pain during treatment will be assessed by the patient using a Visual Analogue Scale (VAS) for pain. The condition of the wound, need for sharp debridement, overall evaluation of the product and safety parameters are assessed by the health care professional treating the patient and the information is collected in the Case Report Form (CRF)

CONTACTS AND LOCATIONS:
Locations (9):
- Sweden (9):
  - Department of Endocrinology Skåne University Hospital Malmö, Malmo, Skåne County
  - Primary Care Center Tunafors, Eskilstuna, Sörmland
  - Wästerläkarna Primary Care Center, Gothenburg, Västra Frölunda
  - Carlanderska Sjukhuset, Gothenburg, Västra Götaland County
  - Medicinkliniken, Diabetescentrum, Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County
  - Närhälsan Olskroken Primary Care Center, Gothenburg, Västra Götaland County
  - Hudmottagningen Skaraborgs Sjukhus, Skövde, Västra Götaland County
  - Dept of Orthopaedic Surgery, Mölndal
  - Sårcentrum Södersjukhuset Stockholm, Stockholm

IPD SHARING:
Plan to Share IPD: No